CLINICAL TRIAL: NCT07343284
Title: Effect of a Nursing Intervention Based on Health Education on Functionality, Depression Symptoms, and Quality of Life in Patients With Ischemic Stroke: A Quasi-Experimental, Longitudinal, and Prospective Clinical Trial
Brief Title: Nursing Health Education to Improve Functionality and Quality of Life After Ischemic Stroke
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Félix Martínez Eiriz, Collaborating Investigator, University of Santiago de Compostela
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025/419
Record Dates: First submitted 2025-12-10; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Ischemia Stroke; Post-stroke Depression; Post-stroke; Quality of Life; Health Education
Keywords: Ischemic stroke; Nursing; Depression; Health education; Quality of life
MeSH Terms: conditions — Ischemic Stroke; Health Education; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological Intervention (Experimental): The educational sessions are based on meaningful learning and incorporate constructivist, cognitive, and behavioral approaches. The program consists of three core components:
  Session 1: Early stroke symptoms and recognition Session 2: Living with stroke: daily care and self-management Session 3: Mood management
  In addition, a workshop (Session 4) will be delivered focusing on depression management through the development of coping strategies, including full-breathing techniques, relaxation exercises, psychotherapy tools, and and mindfulness practices.
  Considering that 35 patients will receive the health education program, an estimated 3-4 groups of 8-12 participants will be formed, each attending the sessions with the same instructor.
  Interventions: Behavioral: Health education Program
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: Health education Program — The program consists of three core components: Session 1: Early stroke symptoms and recognition; Session 2: Living with stroke and daily self-care; and Session 3: Mood management. Additionally, a workshop (Session 4) will be delivered to address depressive symptoms through the development of coping strategies such as full-breathing techniques, relaxation methods, psychotherapy-based exercises, and mindfulness. All sessions will preferably be conducted in group format. Detailed session content is provided in Annex II.
  Considering that 35 patients will receive the health education program, an estimated 3-4 groups of 8-12 participants will be formed, each attending the sessions under the same instructor.
  Schedule
  The sessions will be delivered over two separate days:
  Day 1 (40 minutes):
  Session 1: Early stroke symptoms and their recognition Session 2: Living with stroke: daily care and self-management
  Day 2 (40 minutes):
  Session 3: Mood and depression management Session 4: Relaxa
  Arms: Psychological Intervention

SUMMARY:
This study is titled "Effect of a Nursing Intervention Based on Health Education on Functionality, Depression Symptoms, and Quality of Life in Patients with Ischemic Stroke." It is a quasi-experimental, longitudinal, prospective clinical trial that will beconducted with patients who have suffered an ischemic stroke and were treated in the neurology unit of the Lucus Augusti University Hospital, the same center where this study will take place.

The primary objective of the study is to determine the effect of a nursing intervention based on health education on quality of life and depression symptoms in individuals who have experienced an ischemic stroke.

To achieve this objective, variables such as cognitive status, depression symptoms, autonomy and ability to perform basic activities of daily living, neurological deficits, and quality of life will be assessed.

Regarding the total number of subjects to be studied, according to the Stroke Atlas in Galicia published by the Spanish Society of Neurology in 2018, the autonomous community of Galicia had a population of 2,701,819 inhabitants. Applying an incidence rate of 187.4 cases per 100,000 inhabitants according to the IBERICTUS study, an estimated 5,064 new stroke cases occur each year in Galicia. The province of Lugo had 324,842 inhabitants as of January 1, 2024, according to the INE; therefore, applying the same incidence rate, an estimated 609 new stroke cases occur per year. Considering the proportion of ischemic strokes compared to other types of strokes (80:20), the estimated number of ischemic stroke cases in Lugo would be 487. The representative sample size of stroke patients in the province of Lugo would be 70 patients, with 35 patients receiving the intervention and 35 serving as controls.

Independent Variables:

Sociodemographic: sex, age, event date. Clinical: stroke type, treatment modality (rt-PA or thrombectomy), falls, pain, pressure ulcers, aspiration, pneumonia, dysphagia, vital signs.

Health education: received vs. not received.

Dependent Variables:

Cognitive status (MMSE). Depression symptoms (BDI). Autonomy and ADL performance (Barthel Index). Neurological deficits (NIHSS). Quality of life (European Quality of Life Scale).

Instruments Mini-Mental State Examination (MMSE) Beck Depression Inventory (BDI) Barthel Index NIH Stroke Scale (NIHSS) Visual Analogue Scale (VAS) European Quality of Life Scale (EQLS)

ELIGIBILITY:
Inclusion Criteria:

* Anterior or posterior cerebral occlusion

Exclusion Criteria:

* Intracranial hemorrhage
* Pregnancy
* Cognitive incapacity for participation
* Refusal to participate in the study and administer the questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Depression Symptoms | Baseline, 3 months, and 6 months post-intervention
  Depressive symptoms will be assessed using the Beck Depression Inventory (BDI). This measure evaluates changes in mood and depressive symptomatology in patients who have experienced an ischemic stroke. Scores will be compared between the intervention group (receiving the health education program) and the control group to determine the effect of the nursing-led intervention on depression levels.
Health-Related Quality of Life | Baseline, 3 months, and 6 months post-intervention
  Quality of life will be assessed using the European Quality of Life Scale (EQLS). Comparisons between intervention and control groups will evaluate the effect of the nursing-led health education program on overall well-being and life satisfaction in post
Cognitive Status | 3 months, and 6 months post-intervention
  Cognitive function will be assessed using the Mini-Mental State Examination (MMSE). Scores will be compared between the intervention and control groups to evaluate the effect of the nursing-led health education program on cognitive performance in post-ischemic stroke patients.
Autonomy and Performance in Activities of Daily Living | Baseline, 3 months, and 6 months post-intervention
  Autonomy and the ability to perform basic activities of daily living will be measured using the Barthel Index. The study will compare changes in functional independence between the intervention and control groups.
Neurological Deficit | Baseline, 3 months, and 6 months post-intervention
  Neurological deficits will be assessed using the National Institutes of Health Stroke Scale (NIHSS). Differences between intervention and control groups will be analyzed to determine the impact of the health education program on neurological recovery.

DOCUMENTS (1):
  • Study Protocol (2025-10-22): https://cdn.clinicaltrials.gov/large-docs/84/NCT07343284/Prot_000.pdf